CLINICAL TRIAL: NCT05177822
Title: Interleukin-1 Blockade in Acute Myocardial Infarction to Prevent Heart Failure: The Virginia - Anakinra Remodeling Trial 4
Brief Title: Interleukin-1 Blockade in Acute Myocardial Infarction to Prevent Heart Failure
Acronym: VA-ART4
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HM20022826; R01AG076360 (NIH)
Record Dates: First submitted 2021-12-14; First posted 2022-01-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- anakinra (Experimental)
  Interventions: Drug: Anakinra
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Anakinra — Anakinra 100 mg/0.67 mL daily subcutaneous injection for up to 14 days, including up to 9 days outpatient treatment;
  Other Names: Kineret
  Arms: anakinra
Other: Placebo — 0.9% NaCl/0.67 mL daily subcutaneous injection for up to 14 days, including up to 9 days outpatient treatment.
  Arms: placebo

SUMMARY:
Patients who have a heart attack are at high risk for future development of heart failure ('weakening of the heart'). The researchers believe that the reaction of the heart muscle to injury (inflammation) during a heart attack may be contributing to the risk of heart failure. The current study will test the ability of an anti-inflammatory medicine (anakinra) to block the inflammation in the body during and after a heart attack.

DETAILED DESCRIPTION:
Anakinra (Kineret®) is a 'copy' of a naturally occurring protein made by the body to block inflammation. The US Food and Drug Administration (FDA) has approved anakinra 100 mg daily for the treatment of rheumatoid arthritis but anakinra is not currently approved for the treatment of heart disease. Anakinra is generally well-tolerated, but can cause pain or redness at the injection site and may affect risk of infections. The study team will work with participants to help avoid (or manage) any side effects throughout the study.

The study is designed to measure how well anakinra can protect participants from developing heart failure. Participation in this study will last approximately 1 year. During the first 2 weeks of the study, participants will receive an injection with anakinra or placebo (a liquid that looks like anakinra but contains no active medicine). While hospitalized, a nurse will do the injections for participants; upon discharge participants will be taught to give the remaining injections at home. Assignment to treatment with anakinra or placebo will be determined by randomization (like the "flip of a coin"). Approximately 84 people will participate in this study over the course of 4 years.

ELIGIBILITY:
Inclusion Criteria:

All criteria need to be met.

* Acute ST segment elevation myocardial infarction defined as:

  * chest pain, consistent with angina, within the prior 12 hours (for intermittent pain lasting more than 12 hours, the time from the when the pain became severe and constant);
  * ST segment elevation on ECG >1 mm in 2 or more anatomically contiguous leads;
  * Reperfusion strategy planned or completed (including percutaneous coronary intervention or fibrinolysis)
* Age >21 years.

Exclusion Criteria:

Subjects will not be eligible if they meet any of the following exclusion criteria.

* Pregnancy;
* Inability to obtain consent from patient;
* History of prior STEMI or of systolic heart failure (LVEF<40%);
* Contraindications to treatment with anakinra (i.e. prior allergic reaction to Kineret® or E. coli derived products);
* Duration of chest pain >12 hours at time of coronary artery catheterization (continuously - see exceptions in Inclusion Criteria) or coronary artery intervention >12 hours earlier (see exceptions in Inclusion Criteria)[max duration of chest pain 24 hours];
* Failed reperfusion strategy (unsuccessful percutaneous coronary intervention);
* Need or plan for emergent cardiac surgery;
* Anticipated inability to complete a cardiopulmonary exercise test (CPET) on a treadmill at follow up visit at 42 days (i.e. amputee, wheel-chair bound, severe non-cardiac illness limiting mobility).
* Active infection (such as acute, i.e. COVID-19, or chronic/recurrent infectious disease i.e HBV, HCV, and HIV/AIDS-but excluding HCV+ patients with undetectable plasma RNA)
* Acute or chronic inflammatory disease or immunosuppressive therapies (including oral corticosteroids at a dose of prednisone equivalent of 0.5 mg/kg/day but not including inhaled or low dose oral corticosteroids or non-steroidal anti-inflammatory drugs).
* Neutropenia (<1,500/mm3 or <1,000/mm3 in African-American patients).
* Active acute or chronic psychiatric illness that in the opinion of the investigator may prevent from complying with study instructions;
* Stage V chronic kidney disease (estimated glomerular filtration rate 15 mL/min/1.73m2 or less) or on renal-replacement therapy (a GFR ≥45 mL/min/1.73m2 is required for the cardiac magnetic resonance portion of the study);
* Limited English Proficiency that in the opinion of the investigator may prevent from understanding the content of the informed consent form and instructions during the tests required for the study.
* Any comorbidity limiting survival or ability to complete the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption (peak VO2) | 6 weeks
  Peak VO2 (expressed as % of predicted) will be assess using cardiopulmonary exercise testing (CPET)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Van Tassell, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
A simplified and fully de-identified database will be made available for sharing in accordance with requirements for National Institute on Aging (NIA) data repository datasets and associated documentation for submission to the Biological Specimen and Data Repository Information Coordinating Center (BioLINCC) and the NIA Guidance on Sharing Data and other Resources, within 3 years of completion of the study.